CLINICAL TRIAL: NCT02685839
Title: Development of an Intelligent POWER Rehabilitation Cluster Machine and Its Clinical Testing and Assessment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-06-003B
Record Dates: First submitted 2016-01-05; First posted 2016-02-19 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Frailty Syndrome; Intelligent POWER Rehabilitation Cluster Machine
Keywords: frailty syndrome, Intelligent POWER Rehabilitation Cluster Machine, Internet of Things, wearable
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional rehabilitation (Active Comparator): Each subject will do traditional rehabilitation work two times per week and one hour at a time
  , lasting 24 weeks.
  Interventions: Other: general physical therapy
- Power rehabilitation (Experimental): Each subject will do Power rehabilitation work with motion tracking and biofeedback recording two times per week and one hour at a time, lasting 24 weeks.
  Interventions: Device: Intelligent POWER Rehabilitation Cluster Machine

INTERVENTIONS:
Device: Intelligent POWER Rehabilitation Cluster Machine
  Arms: Power rehabilitation
Other: general physical therapy
  Arms: Traditional rehabilitation

SUMMARY:
Elderly care has become one of the most important subjects in Taiwan and "frailty syndrome" are the most common problems among the elderly. In view of this trend, Taipei Veteran Memorial Hospital imported POWER rehabilitation from Japan in 2008. While showing significant clinical benefits, investigators have found that the system still has certain limitations (e.g. high cost, requires large space, patients must commute to the center, lacks real-time objective feedback , boring routines makes staying power to motivate patients for long term rehabilitation programs.)

To overcome the above limitations, this project proposes an evidence-based rehabilitation model that accounts for actual clinical need and collaborates with our engineering team to develop a "cluster" , "wearable" and "Brain-Computer Interface System" version of POWER rehabilitation system. Combining cloud technology, investigators now introduce internet-of-things into the POWER rehabilitation procedure. The result will lower the burden of clinical support personnel, and provide an opportunity to quantify "frailty syndromes" so as to allow objective and quantitative scientific evaluation, leading to a more objective clinical diagnosis.

In addition, this project further proposes a virtual-reality (VR) system for POWER rehabilitation, as well as designs for the VR sceneries. Through the use of different animated 3D VR sceneries and interactive game design, investigators can make rehabilitation interesting and fun for the patients, motivating long-term compliance of the patients, thereby, improving the clinical outcome of POWER rehabilitation.

This project has the potential to create an innovative solution to address the current bottlenecks of our rehabilitation treatment model. Successful development of the system will offer rehabilitation clinicians more treatment options, lower the cost of supporting staff, reduce commuting cost for the patients, and elevate patient desire to comply with the treatment program. Finally, the system will not only enhance Taiwan's academic reputation in the international arena, it will also generate new commercial opportunities for Taiwan and contribute to Taiwan economic development.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 to 85
* Cardiovascular Health Study (CHS) frailty criteria
* willing to sign agreement

Exclusion Criteria:

* fracture w/o healing
* severe joint injury
* acute stroke or myocardial infarction (< 3 months)
* cardiac arrhythmia / unstable blood pressure
* disorientation or intellectual deterioration
* muscle contracture deformity
* pregnancy

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Tilburg Frailty Indicator (TFI) | Changes from baseline in physical examination at 12, 16 weeks
  The TFI contains two parts, sociodemographic questions including questions on multimorbidity, lifestyle, life events and living environment (part A) and the assessment of components of frailty (part B). Frailty is assessed with 15 items divided into physical, social and psychological domains. All item scores are summed into a frailty score ranging from 0-15. Persons with a total TFI score ≧5 are considered to be frail.

SECONDARY OUTCOMES:
balance test (sec) | Changes from baseline in physical examination at 12, 16 weeks
  single leg stance with eyes open
flexibility test_1st (cm) | Changes from baseline in physical examination at 12, 16 weeks
  truck flexion test in standing position
flexibility test_2nd (cm) | Changes from baseline in physical examination at 12, 16 weeks
  truck flexion test in sitting position
general mobility test (sec) | Changes from baseline in physical examination at 12, 16 weeks
  timed up and go test
hand-eye coordination test (sec) | Changes from baseline in physical examination at 12, 16 weeks
  grasp an falling rod
muscle endurance test (times/2 min) | Changes from baseline in physical examination at 12, 16 weeks
  step in place with hip raising to level
muscle strength test (kgw) | Changes from baseline in physical examination at 12, 16 weeks
  grip strength
visual test | Changes from baseline in physical examination at 12, 16 weeks
  traditional visual test in the letter C
hearing test (sec) | Changes from baseline in physical examination at 12, 16 weeks
  traditional hearing test with high frequency(4096Hz) and low frequency(512Hz) tuning fork
Activity of daily living (ADL) | Changes from baseline in ADL at 12, 16 weeks
  This index measures the extent to which somebody can function independently and has bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. The index also indicates the need for assistance in care. Scores range from 0 to 100 with higher scores indicating greater independence.
Instrumental Activities of Daily Living (IADL) | Changes from baseline in physical examination at 12, 16 weeks
  IADL's are activities related to independent living and include preparing meals, managing money, shopping for groceries or personal items, performing light or heavy housework, doing laundry, and using a telephone. The total score may range from 0 - 8. A lower score indicates a higher level of dependence.
Functional Independence Measure (FIM) | Changes from baseline in physical examination at 12, 16 weeks
  The Functional Independence Measure (FIM) scale assesses physical and cognitive disability. This scale focuses on the level of disability indicating the burden of caring for them. The scale includes 18 items. Each item is scored from 1 to 7 based on level of independence, where 1 represents total dependence and 7 indicates complete independence. Possible scores range from 18 to 126, with higher scores indicating more independence.
36-Item Short Form Health Survey (SF-36) | Changes from baseline in physical examination at 12, 16 weeks
  The SF-36 consists of eight sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Si Huei Lee, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Power Rehabilitation Room, Taipei Veterans General Hospital Integrative Rehabilitation Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pialoux T, Goyard J, Lesourd B. Screening tools for frailty in primary health care: a systematic review. Geriatr Gerontol Int. 2012 Apr;12(2):189-97. doi: 10.1111/j.1447-0594.2011.00797.x. Epub 2012 Jan 10. PMID 22233158
- [Background] Fung J, Richards CL, Malouin F, McFadyen BJ, Lamontagne A. A treadmill and motion coupled virtual reality system for gait training post-stroke. Cyberpsychol Behav. 2006 Apr;9(2):157-62. doi: 10.1089/cpb.2006.9.157. PMID 16640470
- [Background] Eriksson L, Lindstrom B, Ekenberg L. Patients' experiences of telerehabilitation at home after shoulder joint replacement. J Telemed Telecare. 2011;17(1):25-30. doi: 10.1258/jtt.2010.100317. Epub 2010 Nov 12. PMID 21075802
- [Background] Cherney LR, van Vuuren S. Telerehabilitation, virtual therapists, and acquired neurologic speech and language disorders. Semin Speech Lang. 2012 Aug;33(3):243-57. doi: 10.1055/s-0032-1320044. Epub 2012 Jul 31. PMID 22851346
- [Background] Sharma S, Ward EC, Burns C, Theodoros D, Russell T. Training the allied health assistant for the telerehabilitation assessment of dysphagia. J Telemed Telecare. 2012 Jul;18(5):287-91. doi: 10.1258/jtt.2012.111202. Epub 2012 Jul 11. PMID 22790011
- Available data/document: Clinical Study Report — http://goo.gl/FilVtL